CLINICAL TRIAL: NCT01132768
Title: Effects of Angiotensin-Receptor Blockade With Olmesartan on Carotid Atherosclerosis in Patients With Hypertension: The Confirmatory Olmesartan Plaque Regression Study
Brief Title: The Confirmatory Olmesartan Plaque Regression Study
Acronym: CONFIRM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSE-OLM-01-09
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2012-03

CONDITIONS: Essential Hypertension; Carotid Plaque
MeSH Terms: conditions — Essential Hypertension | interventions — Atenolol; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atenolol (Active Comparator): Atenolol (ATE) 50 mg and/or 100 mg tablets, oral, once daily.
  Interventions: Drug: Atenolol
- Olmesartan medoxomil (Experimental): Olmesartan medoxomil (OM), 20 mg and/or 40 mg, oral, once daily.
  Interventions: Drug: olmesartan medoxomil

INTERVENTIONS:
Drug: Atenolol — Atenolol (ATE) 50 mg and/or 100 mg tablets, oral, once daily
  Arms: Atenolol
Drug: olmesartan medoxomil — Olmesartan medoxomil (OM), 20 mg and/or 40 mg, oral, once daily
  Arms: Olmesartan medoxomil

SUMMARY:
Effect of olmesartan medoxomil (20-40 mg) on plaque regression in hypertensive patients with carotid atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Caucasian outpatients aged > 40 years.
* High BP defined as mean SeSBP/SeDBP ≥ 140/90 mmHg.
* One or more of the following additional risk factors:
* Smoking;
* Dyslipidaemia (high-density lipoprotein (HDL)-cholesterol < 0.9 mmol/L or low-density lipoprotein (LDL)-cholesterol > 2.6 mmol/L, or triglycerides > 1.7 mmol/L);
* Left ventricular hypertrophy;
* Cardio-cerebrovascular events > 6 months ago;
* Presence of target organ damage.
* Non-calcified (not marked shadowing) plaque in the CC artery, in the internal carotid artery or the carotid bulb with a PV ≥ 0.040 cm³ (≥ 40 µL) according to the measurements of EUTARC.

Exclusion Criteria:

* Secondary or high grade hypertension including grade III hypertension (SeSBP of > 180 mmHg or SeDBP of > 105 mmHg).
* Stroke, myocardial infarction within the previous 6 months.
* Interventional or surgical vascular treatment within the previous 3 months.
* Presence of significant narrowing of the aortic or bicuspid valve and severe obstruction of cardiac outflow (hypertrophic cardiomyopathy).
* Symptomatic heart failure.
* Diabetes.
* Chronic obstructive pulmonary disease (COPD) or asthma.
* Claudication intermittens stage II b or higher.
* Clinical evidence of severe renal disease [including renovascular occlusive disease, nephrectomy and/or renal transplant, creatinine clearance of < 30 mL/min, macroalbuminuria (> 300 mg albumin/24 hours or 300 µg albumin/mg creatinine)].
* Treatment with angiotensin converting enzyme (ACE)-inhibitors or angiotensin-receptor blockers (ARBs) during last 3 months.
* Start of treatment with a lipid-lowering agent or modification of dosage within last 3 months.
* Electrocardiographic (ECG) evidence of 2nd or 3rd degree atrioventricular (AV) block, atrial fibrillation, cardiac arrhythmia (requiring therapy) or bradycardia (< 50 beats/min at rest).
* Known intolerance to study drugs.
* Impaired liver function tests suggesting severe liver disorder.
* Any life threatening disease.
* Duplex sonographically determined stenosis of the common or internal carotid artery > 75%.
* Plaque with marked shadowing from calcification.
* Target plaques in CC artery extending into both internal and external arteries.
* Pregnant or lactating female subjects.
* Female subjects of childbearing potential without adequate contraception: intra-uterine devices, hormonal contraceptives, either oral, depot, patch or injectable and double barrier methods such as condoms or diaphragms with spermicidal gel or foam. If a female becomes pregnant during the trial, she has to be withdrawn immediately (see section 9.4).
* Subject is currently enrolled in or has not yet completed at least 30 days since ending another investigational device or drug study or is receiving other investigational agents.
* Subject has previously entered this study.
* Subjects who have received ATE within 30 days prior to entering the active treatment phase.
* Subjects who are unwilling or unable to provide informed consent or to participate satisfactorily for the entire trial period.
* Subjects with history of alcohol and or drug abuse.
* Subjects with known malabsorption syndrome.
* Subjects who had donated or lost 450 mL or more blood during the last three months before Screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in carotid plaque volume | 78 weeks (week 78 - week 0)
  change in carotid plaque volume (PV) from baseline (week 0) as assessed by 3-D ultrasonography after 78 weeks of double-blind treatment with Olmesartan (OM) 20-40 mg daily compared to Atenololo (ATE) 50-100 mg daily (week 78 - week 0).

SECONDARY OUTCOMES:
Change in plaque volume after 52 weeks, olmesartan versus atenolol | 52 weeks (week 52 - week 0)
  change in plaque volume PV from baseline (week 0) to Week 52 on olmesartan therapy versus atenolol therapy
Percentage changes of PV from baseline to Week 52 for olmesartan versus atenolol. | 52 weeks (week 52-week 0)
  Determine the percentage changes of PV from baseline (week 0) to Week 52 for olmesartan versus atenolol.
Percentage changes of PV from baseline to Week 78 for olmesartan versus atenolol. | 78 weeks (week 78 - week 0)
  Determine the percentage changes of PV from baseline (Week 0) to Week 78 for olmesartan versus atenolol.
Change in seated diastolic blood pressure (SeDBP) from baseline to Week 52 for olmesartan versus atenolol. | 52 weeks (week 52 - week 0)
  Determine the change in seated diastolic blood pressure (SeDBP) from baseline (week 0) to Week 52 for olmesartan versus atenolol.
Change in seated diastolic blood pressure (SeDBP) from baseline to Week 78 for olmesartan versus atenolol. | 78 weeks (week 78 - week 0)
  Determine the change in seated diastolic blood pressure (SeDBP) from baseline (week 0) to Week 78 for olmesartan versus atenolol.
Change in seated systolic blood pressure (SeSBP) from baseline to Week 52 for olmesartan versus atenolol. | 52 weeks (week 52 - week 0)
  Determine the change in seated systolic blood pressure (SeSBP) from baseline (week 0)to Week 52 for olmesartan versus atenolol.
Change in seated systolic blood pressure (SeSBP) from baseline to Week 78 for olmesartan versus atenolol. | 78 weeks (week 78 - week 0)
  Determine the change in seated systolic blood pressure (SeSBP) from baseline (week 0) to Week 78 for olmesartan versus atenolol.
Change in PV from baseline to Week 52 after adjustments for changes in SeDBP from baseline. | 52 weeks (week 52 - week 0)
  Determine the change in PV from baseline (week 0) to Week 52 after adjustments for changes in SeDBP from baseline.
Change in PV from baseline to Week 78 after adjustments for changes in SeDBP from baseline. | 78 weeks (Week 78 - week 0)
  Determine the change in PV from baseline (week 0) to Week 78 after adjustments for changes in SeDBP from baseline.
Change in PV from baseline to Week 52 after adjustments for changes in SeSBP from baseline. | 52 weeks (week 52 - week 0)
  Determine the change in PV from baseline (week 0) to Week 52 after adjustments for changes in SeSBP from baseline.
Change in PV from baseline to Week 78 after adjustments for changes in SeSBP from baseline. | 78 weeks (Week 78- week 0)
  Determine the change in PV from baseline (week 0) to Week 78 after adjustments for changes in SeSBP from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus O Stumpe, MD, Principal Investigator — Centre of Preventative Medicine
Locations (1):
- Sesto Fiorentino, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/